CLINICAL TRIAL: NCT07104357
Title: The Effect of Inspiratory Muscle Training on Dysfunctional Breathing and Functional Ability in Patients With Chronic Heart Failure. A Study Protocol for a Randomized Controlled Trial
Brief Title: The Effect of Inspiratory Muscle Training on Breathing Pattern and Functionality in Patients With Chronic Heart Failure.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Georgios Mitsiou, Laboratory Teaching Staff, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 51604/04-06-2025
Record Dates: First submitted 2025-07-07; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Breathing Pattern Disorder
Keywords: inspiratory muscle training; dysfunctional breathing; functional ability; chronic heart failure

STUDY DESIGN:
Intervention Model Description: This single-center, randomized controlled, single-blinded clinical trial is designed to investigate the effectiveness of inspiratory muscle training on breathing pattern and functional ability in patients with chronic heart failure
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized controlled trial (Experimental): The intervention group will be trained with inspiratory muscle training for 4 weeks. Inspiratory Muscle Training has been designed to enhance respiratory muscle function through targeted exercises, to strengthen the respiratory muscles, ,thereby improving overall respiratory efficiency
  Interventions: Device: Inspiratory muscle training
- Control group (No Intervention): The control group will receive standard care

INTERVENTIONS:
Device: Inspiratory muscle training — Participants will perform 20 sessions of respiratory muscle strengthening (20 minutes at 30-60% of MIP), using the Threshold Inspiratory Muscle Training device
  Arms: Randomized controlled trial

SUMMARY:
The effect of inspiratory muscle training on breathing pattern and functionality in patients with chronic heart failure.

DETAILED DESCRIPTION:
The study protocol aims to examine the impact of inspiratory muscle training on dysfunctional breathing and functional ability in patients with chronic heart failure. Inspiratory muscle training is a low-cost intervention that might improve the breathing pattern, functionality and overall quality of life in patients with chronic heart failure

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≥ 18 years
* diagnosis of heart failure within the previous three to twelve months
* current outpatients in a stable optimal medical regimen for at least 3 months
* able to perform inspiratory muscle training
* clinically stable, without hospital admission in the previous 3 months and without participation in any other training program in the previous 6 months

Exclusion Criteria

* unstable angina
* recent acute myocardial infarction
* uncontrolled hypertension
* valve disease
* peripheral arterial disease
* 6MWT assessment of less than 300 meters
* previous pulmonary disease (forced vital capacity <80% of predicted and/or forced expiratory volume in 1 s <70% of predicted)
* history of exercise-induced asthma
* smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic Thickness | From enrollment to the end of treatment at 4 weeks
  Diaphragmatic thickness measured by ultrasound is a non-invasive, widely used method to assess diaphragm structure in patients with chronic heart failure. Thickness is measured between the pleural and peritoneal lines at end-expiration and end-inspiration
Dysfunctional breathing | From enrollment to the end of treatment at 4 weeks
  Dysfunctional breathing refers to abnormal breathing patterns that are often related to the heart's inability to supply blood effectively, affecting respiratory function. Dysfunctional breathing will be assessed with the Hi-Lo breathing test, an observational clinical test used to assess breathing pattern and diaphragm function. The clinician observes and palpates whether the movement is greater under the upper chest hand (Hi) or lower abdomen hand (Lo).The test is scored as "Yes" if upper chest (apical) breathing predominates and "No" if normal diaphragmatic breathing is present.
Functional ability | From enrollment to the end of treatment at 4 weeks
  Functional ability refers to how well patients can perform daily activities and maintain independence despite their cardiac condition. It will be assessed with the 6-Minute Walk Test (6MWT), a simple and effective tool that evaluates the maximum distance a person can walk in six minutes. The outcome reflects the integrated response of the cardiovascular system mainly, and exercise tolerance.

SECONDARY OUTCOMES:
Maximal inspiratory pressure | From enrollment to the end of treatment at 4 weeks
  It is a measure of the strength of inspiratory muscles, primarily the diaphragm. MIP is a reliable and reproducible measure that does not depend on the patient's respiratory flow.
Functional Dyspnea | From enrollment to the end of treatment at 4 weeks
  Functional dyspnea will be measured with the Medical Research Council (MRC) Dyspnea scale, a simple grading system to evaluate the functional disability due to dyspnea. The scale ranges from 1 to 5, where 1 indicates breathlessness only with strenuous exercise and 5 indicates breathlessness that prevents leaving the house or occurs when dressing or undressing. Higher scores represent worse functional status (more severe dyspnea).
Health Related Quality of life | From enrollment to the end of treatment at 4 weeks
  Quality of life will be evaluated with the Short Form Survey, a questionnaire with 12-items, that measures quality of life in terms of physical and mental health. It generates scores typically ranging from 0 to 100, with higher scores indicating better health status and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Irini Grammatopoulou, Phd, Post Doc, Study Director — University of West Attica, Athens, Greece

IPD SHARING:
Plan to Share IPD: No